CLINICAL TRIAL: NCT02610387
Title: The Effects of tDCS Combined With Balance Training on Lower Limbs Spasticity in Chronic Stroke Patients ( A Randomized Controlled Trial)
Brief Title: The Effects of tDCS Combined With Balance Training on Lower Limbs Spasticity in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fariba Yadolahi, MD-MPH-PhD candidate, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS and Spasticity
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Ischemic Stroke
Keywords: tDCS; stroke; Spasticity
MeSH Terms: conditions — Ischemic Stroke; Stroke; Muscle Spasticity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1:tDCS (Active Comparator): Transcranial direct current stimulation (tDCS) Participants underwent tDCS(2mA) brain stimulation (20 minutes) and simultaneous balance training(20 minutes) for 5 consecutive days
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Arm 2: Sham tDCS (Sham Comparator): Sham tDCS and simultaneous balance training(20 minutes) for 5 consecutive days
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Participants underwent tDCS(2mA) brain stimulation for 20 minutes plus balance training for 20 minutes for 5 consecutive days.
  Arms: Arm 1:tDCS
Device: Sham tDCS — During sham stimulation, the current ramped up for 30 seconds, ramped back down for 30 seconds, and then remained off for the duration of the stimulation plus balance training for 20 minutes for 5 consecutive days.
  Arms: Arm 2: Sham tDCS

SUMMARY:
Spasticity is one of the most common disorders in patients with central nervous system diseases such as stroke. Transcranial direct current stimulation stimulation (tDCS) is a noninvasive tool that can be used to modulate cortical excitability of the leg motor area, and the spinal motor circuits as well.

Objective:The objectives of this study is to examine the efficacy of anodal tDCS combined with Biodex balance training on lower limbs spasticity in chronic stroke patients using laboratory and clinical assessments.

DETAILED DESCRIPTION:
In a randomized, sham-controlled, double-blinded clinical study, hemiplegic chronic stroke patients are randomized to receive active tDCS delivered to lesioned leg motor cortex (CZ) or sham combined with balance training with Biodex balance system.

Experimental group receive tDCS stimulation (2mA) for 20 min, 5 sessions in five days paired with 20 min balance training.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* first-ever ischemic stroke;
* chronic phase of recovery (>6 months);
* ability to walk 6- meter supported or unsupported;
* ability to stand at least unsupported for 40-seconds with eyes closed;
* only ischemic stroke involving middle cerebral artery (MCA) territory confirmed by CT or MRI.

Exclusion Criteria:

* Use of any neuro- or psycho-active medications that alters balance;
* any other neurological conditions or sensory disorders affecting postural control; such as brain tumor, or substance abuse; orthopedic diseases;
* ongoing/recent (within 3 months) balance rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09-12; Primary Completion 2017-12-20 (Estimated); Study Completion 2017-12-20 (Estimated)

PRIMARY OUTCOMES:
Spasticity (Modified Ashworth scale) | After 5 days
  Modified Ashworth scale(MAS)

SECONDARY OUTCOMES:
Motoneuron excitability (H-reflex latency) | After 5 days
  H-reflex latency
Motoneuron excitability | After 5 days
  H Max/M MaxRatio

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti Univesity of Medical sciences, Tehran, Velenjak, Iran